CLINICAL TRIAL: NCT01180231
Title: Assessment of the Effect of Moxonidine and Diet on Cardiac, Renal and Endothelial Function in Young Subjects With Abdominal Obesity
Brief Title: Study of the Effect of Moxonidine and Diet on Sympathetic Functions in Young Adults With Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Dr Elisabeth Lambert, BakerIDI Heart and Diabetes Institute
Allocation: Non-Randomized | Masking: Single
Other Study IDs: Project 168-10
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Obesity; Overweight
Keywords: Overweight or obese young adults (18 to 30 years old) with no previous history of cardiovascular disease/psychiatric illness, and not on medications
MeSH Terms: conditions — Obesity; Overweight; Mental Disorders | interventions — moxonidine; Diet Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Moxonidine (Active Comparator)
  Interventions: Drug: Moxonidine (Physiotens)
- Diet (Active Comparator)
  Interventions: Other: Dietary intervention
- Moxonidine and diet (Active Comparator): Subjects will be asked to take moxonidine and follow dietary plan designed by a qualified nutritionist for 6 months.
  Interventions: Drug: Moxonidine (Physiotens); Other: Dietary intervention
- Control (No Intervention): Subjects will not be asked to take any interventions.

INTERVENTIONS:
Drug: Moxonidine (Physiotens) — Subjects will be asked to take moxonidine, dosage to be determined prior to commencement by a medical doctor for 6 months duration.
  Other Names: Physiotens
  Arms: Moxonidine; Moxonidine and diet
Other: Dietary intervention — Subjects will be asked to follow dietary plans designed by a qualified nutritionist for 6 months.
  Arms: Diet; Moxonidine and diet

SUMMARY:
The prevalence of obesity is increasing rapidly among adults and has more than doubled in the past 10 years. The metabolic syndrome (MS) is often associated with obesity. It is characterized by abdominal obesity, high blood pressure, unfavorable blood cholesterol profile, elevated blood sugar and impaired insulin action. Persons with the MS have an increased risk of developing type 2 diabetes as well as heart and kidney disease.

The prevalence of obesity and MS is also very high in children and young adults. While there are increasing numbers of studies assessing risk factors for cardiovascular and kidney disease in middle aged to older obese subjects, few studies have addressed the issue of the presence of obesity in young adults and its association with MS on early damage to the organs such as the kidneys, the heart and the blood vessels. The investigators' laboratory has a particular interest on the sympathetic nervous system, which is an important regulatory mechanism of both metabolic and cardiovascular function, as altered sympathetic activity may play a role in the complications of obesity.

Moxonidine is a medication that is approved in Australia by the Therapeutic Goods Administration to treat high blood pressure. It works by decreasing the activity of the sympathetic nervous system. With the elevation of the sympathetic activity in obesity, the investigators believe moxonidine may have a favourable role in rescuing early organ damage associated with obesity. This study will assess whether treating obese subjects with moxonidine have positive effects on blood vessels, cardiac and kidney function and anxiety disorder. The investigators will also examine the influence of the sympathetic nervous system activity in these possible altered cardiac, kidney and vessel functions.

ELIGIBILITY:
Inclusion Criteria:

* Males age between 18 to 30 years old
* Abdominal obesity according to International Diabetes Federation (IDF) definition

Exclusion Criteria:

* Any medications
* history of cardiovascular disease
* history of diabetes
* history of psychiatric illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
To determine whether moxonidine is able to reverse the early organ damage compared to the effect of weight loss alone, and whether the addition of moxonidine during a weight loss program confers greater beneficial effect.

CONTACTS AND LOCATIONS:
Locations (1):
- BakerIDI Heart and Diabetes Institute, Prahran, Victoria, Australia

REFERENCES:
- [Derived] Lambert EA, Sari CI, Eikelis N, Phillips SE, Grima M, Straznicky NE, Dixon JB, Esler M, Schlaich MP, Head GA, Lambert GW. Effects of Moxonidine and Low-Calorie Diet: Cardiometabolic Benefits from Combination of Both Therapies. Obesity (Silver Spring). 2017 Nov;25(11):1894-1902. doi: 10.1002/oby.21962. Epub 2017 Sep 2. PMID 28865109